CLINICAL TRIAL: NCT05946447
Title: Intra- and Interrater Reliability of Quantitative Ultrasound Assessment of Gastric Content in Term Parturients Before Elective Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-02
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy; Respiratory Aspiration of Gastric Content
Keywords: Gastric Ultrasound
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric Ultrasound (Experimental): Ultrasound measurements of the antrum will be recorded.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — The gastric antrum will be scanned using ultrasound.
  Other Names: Gastric Ultrasound

SUMMARY:
The presence of solid food or fluid residue in the stomach is always a major concern when patients require medical procedures under sedation or general anesthesia, due to the high risk of pulmonary aspiration of the stomach contents. This is especially important in emergency procedures, when a fasting period could not be observed. Pulmonary aspiration of gastric content is a serious perioperative complication of obstetric anesthesia, and it is associated with morbidity and mortality. Information from a bedside ultrasound assessment of the stomach may be a very useful resource to decide whether it's safe to proceed, cancel or delay a surgical procedure. The ultrasound assessment of the stomach content has shown to be very feasible and practical in non-pregnant patients. However, it has not been determined whether the competence reached by anesthesiologists in non-pregnant subjects can be transferred to the obstetric population, especially in term pregnant patients where it could be difficult to identify the stomach because of the presence of the gravid uterus. Although quantitative assessment of the gastric antrum cross-sectional area in terms of intra- and interrater reliability has been evaluated in non-pregnant adults, it remains to be evaluated in pregnant patients. Furthermore, it has not been determined whether the performance of novice operators is comparable to expert operators in the gastric quantitative assessment. This study aims to determine whether trained anesthesiologists can reliably assess the stomach content of pregnant patients by ultrasound, evaluating the inter- and intra-rater reliability of quantitative gastric ultrasound in term pregnant patients comparing anesthesiologists of different level of expertise. The investigators hypothesize a substantial to almost perfect agreement in the intra- and interrater reliability of the antral cross-sectional area among raters in term pregnant patients scheduled for elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* non-laboring term pregnant women scheduled for cesarean delivery under neuraxial anesthesia
* ≥37 weeks gestational age
* ≥18 years of age
* ASA physical status II-III
* weight 50 to 120 kg
* height ≥150 cm
* ability to understand the rationale of the study evaluations.

Exclusion Criteria:

* multiple pregnancy
* known (reported by the study subject) anomalous anatomy of the upper gastrointestinal tract
* previous surgical procedures on the esophagus, stomach or upper abdomen
* patients not following our institutional fasting instructions (8 hours after a meal and 2 hours for clear liquids)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Antral cross-sectional area (supine position) | 5 minutes
  The cross-sectional area (in centimeters squared) of the antrum will be measured with the patient in supine position, using the ultrasound machine. Measurements will be done 3 times, by 2 investigators.
Antral cross-sectional area (right lateral decubitus) | 5 minutes
  The cross-sectional area (in centimeters squared) of the antrum will be measured with the patient in right lateral decubitus position, using the ultrasound machine. Measurements will be done 3 times, by 2 investigators.

SECONDARY OUTCOMES:
Intra-rater reliability calculation | 5 minutes
  Intra-rater reliability will be calculated using the 3 measurements, for each rater.
Inter-rater reliability calculation | 5 minutes
  Inter-rater reliability will be calculated using the 3 measurements, between raters.
Grading of stomach contents | 5 minutes
  Grading scale: grade 0 means no gastric contents are visualized in supine and the right lateral decubitus, grade 1 means gastric contents are visualized in right lateral decubitus but not in supine decubitus, and grade 2 means gastric contents are visualized in both positions
Gastric volume (supine position) | 5 minutes
  Gastric volume (ml) will be estimated using the antral cross-sectional area obtained with the patient in supine position
Gastric volume (right lateral decubitus) | 5 minutes
  Gastric volume (ml) will be estimated using the antral cross-sectional area obtained with the patient in right lateral decubitus.

CONTACTS AND LOCATIONS:
Overall Officials: Cristian Arzola, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada